CLINICAL TRIAL: NCT04847869
Title: Near-Infrared Light Photobiomodulation Treatment for Retinal Vein Occlusion Macular Oedema
Acronym: NIRVO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Responsible Party: Principal Investigator, Elisa Cornish, Dr, University of Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIRVO
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Macula Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Intervention Model Description: 7 eyes with branch retinal vein occlusion, 7 with central retinal vein occlusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIR laser treatment 200mW/cm2 dose (Experimental): Each NIR light treatment will consist of a 90 second exposure of the macula of the study eye to the Ellex Integre NIR laser with the patient fixating on the central aiming beam. The laser light beam is 4.5mm in diameter with a central masked area of 1.0 mm diameter containing the central fixation target. In this way the central macula will be spared in the event of an adverse effect of the laser, which we do not anticipate.
  The patient will be seated at the slit lamp laser delivery system and after the eye has been dilated and anesthetised with topical eye drops a standard fundus contact lens will be placed on the eye through which the post area pole will be visualised while the treatment is delivered. There will be 12 treatments administered over a 5 week period.
  Interventions: Device: Ellex Integre NIR laser

INTERVENTIONS:
Device: Ellex Integre NIR laser — The Ellex Integre NIR (near Infrared Light) Laser dose of 200 mW/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.

SUMMARY:
This pilot study aims to establish that treatment with near infrared light (NIR) reduces cystic macular oedema in patients with a retinal vein occlusion.

DETAILED DESCRIPTION:
Intraocular injections of Vascular Endothelial Growth Factor (VEGF) inhibitors have been shown to improve swelling of central retina (macular oedema) and vision in patients with retinal vein occlusions (RVO), however this treatment comes with potentially sight threatening risks. A less invasive treatment might have many advantages. We recently showed that eyes with macular oedema caused by diabetes, the other main cause of macular oedema, who received treatment with near-infrared (NIR) light was not only safe but was also effective in reducing the swelling. The US Diabetic Retinopathy Research Collaboration are currently recruiting for a larger study of NIR light which may or may not confirm our findings. We propose to test the safety and efficacy of the same NIR light in patients with macular oedema from retinal vein occlusions. We anticipate this may reduce the need for injections of VEGF inhibitors in eyes with RVO, in particular eyes with good vision. This pilot study will help determine whether PBM with NIR for RVO warrants further investigation in a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis macular edema secondary to branch or central vein occlusion (BRVO or CRVO)
* CMT of >300 µm and less than 550 µm;
* Best corrected visual acuity of 6/6 to 6/24 (letters 87 - 53);
* Intraocular pressure < 25 mmHg;
* Written informed consent has been obtained.

Exclusion Criteria:

* Loss of vision due to other causes (e.g. age-related macular degeneration, myopic macular degeneration, DME);
* Known allergy to agents used in the study e.g. fluorescein;
* Women who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using reliable means of contraception;
* Only eye (vision in other eye <6/60);
* Study eye is an amblyopic eye;
* Macular oedema due to other causes;
* Significant diabetic retinopathy;
* An ocular condition that would prevent visual acuity improvement despite resolution of oedema (such as foveal atrophy or substantial premacular fibrosis;
* Previous treatment with any anti-VEGF therapy or investigational drugs in the study eye at any time prior to baseline.
* Previous use of intraocular or periocular steroids in study eye at any time prior to baseline;
* Cataract surgery within the last 3 months;
* Retinal laser treatment within the last 6 months;
* Media opacity including cataract that already precludes adequate macular photography or cataract that is likely to require surgery within 6 months;
* Intercurrent severe disease such as septicaemia, any condition which would affect follow-up;
* History of chronic renal failure requiring dialysis or renal transplant;
* Blood pressure >180/120;
* Participant has a condition or is in a situation that in the investigator's opinion may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in central macular thickness (CMT) measured by optical coherence tomography (OCT) 12 weeks from baseline, in participants with macular edema from a retinal vein occlusion (RVO) | 12 weeks

SECONDARY OUTCOMES:
Reduction in CMT measured by OCT at 5 and 12 weeks from baseline | 5 & 12 weeks
Mean change in vision from baseline | 12 weeks
Percentage of eyes with no central macular edema at 12 weeks | 12 weeks
Percentage of eyes that require rescue treatment | baseline to 12 weeks
  Rescue treatment - intravitreal anti-VEGF
Mean time to rescue treatment | Upto 12 weeks
If rescue treatment required, mean time till next anti-VEGF using prn regimen review | 6 months
Mean time to oedema recurrence (defined as needing intravitreal treatment) if macular edema resolves | 6 months
Changes to deep vascular OCT-Angiography | 12 weeks
Fundus Fluorescein Angiography assessment of leak and capillary closure before (at baseline) and at 12 weeks post baseline after intervention | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elisa E Cornish, MBBS PhD, Principal Investigator — University of Sydney
Locations (1):
- Macular Research Group, Save Sight Institute, The University of Sydney, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792